CLINICAL TRIAL: NCT05586594
Title: Identifying Maturity-onset Diabetes of the Young in Susceptible Emirati Patients Who Are Currently Treated as Type 1 or Type 2 Diabetes Mellitus
Brief Title: Identifying Maturity-onset Diabetes of the Young in Emirati Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Dr Adnan Agha, Assistant Professor, Internal Medicine, College of Medicine and Health Sciences, United Arab Emirates University, United Arab Emirates University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UAEU_CMHS_TWM_IM_MODY_2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Maturity-onset Diabetes of the Young; Monogenic Diabetes; MODY
Keywords: Maturity-onset Diabetes of the Young (MODY); Diabetes Mellitus; Diagnosis; Precision Medicine
MeSH Terms: conditions — Mason-Type Diabetes; Diabetes Mellitus, Type 2; Diabetes Mellitus; Disease | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients labelled as Type 1 or Type 2 Diabetes (Other): paediatric or adult patients already diagnosed with either type 1 or type 2 diabetes mellitus, following up with Tawam Hospital Diabetes clinics for at least 1 year, (who have negative autoimmunity, lack of significant ketosis and either family history of diabetes in one parent or BMI<40).
  Patient with age > 11; both male or female, Emirati patients only, who attended Diabetes clinic Tawam hospital during the last 1 year AND Diagnosed to have Type 1 or Type 2 Diabetes Mellitus diagnosed before the age of 40 and after the age of 6 months (to exclude neonatal diabetes).
  • .
  Interventions: Diagnostic Test: Genetic testing for 4 MODY genes (GCK, HNF1A, HNF4A, HNF1B)

INTERVENTIONS:
Diagnostic Test: Genetic testing for 4 MODY genes (GCK, HNF1A, HNF4A, HNF1B) — Genetic testing for 4 MODY genes (GCK, HNF1A, HNF4A, HNF1B) to look for common non-syndromic MODY in Emirati population

SUMMARY:
Diabetes Mellitus is a disease that affects nearly 1 in 5 people in United Arab Emirates and is one of leading causes of death and disability. The main reason for this condition is either relative or near complete deficiency of essential hormone made by our pancreas called "insulin", which is required to utilize blood sugar (glucose), and insulin shortage leads to increased blood glucose. The common types of this condition include type 2 Diabetes Mellitus (the most common with almost 90% of all diabetes patients having this condition), which is related to mismatch of body requirements and production of essential hormone called insulin (relative deficiency) and type 1 diabetes, in which body's own defense system causes of destruction of insulin producing cells in the pancreas (near complete deficiency of insulin). However, in younger age group (below the age of 35) there is another type of diabetes which affects nearly 1 out 1000 people and is Maturity onset diabetes of the young (MODY). MODY is a condition passed by parents in 50% of the kids due to an affected single gene and most common forms of MODY do not require any Insulin treatment. However as type 1 Diabetes is generally identified in younger age group, 80% of patient who have MODY cannot be diagnosed and are labelled with other forms of diabetes instead, and may receive unnecessary insulin injections. Although, there has been a lot of research done in the west on prevalence of MODY in white/Caucasian population, the studies in Middle East are minimal. Also, in the white/Caucasian population, a reliable risk calculator has been developed that predicts the risk of having MODY, which if found to be high, is then confirmed by genetic testing for MODY. There is no study available on presence of MODY or on the reliability of the MODY risk calculator among young Emirati population. There is also no data on MODY being misdiagnosed as other forms of diabetes in Emirati population.

This study proposal aims to address this gap of knowledge and assess the reliability of MODY calculator in young Emirati patients with diabetes and to see if any MODY patient exist in Diabetes clinics of Tawam hospital Abu Dhabi, who may have been misdiagnosed as type 1 or type 2.

DETAILED DESCRIPTION:
Background:

Diabetes Mellitus (DM) affects more than half a billion people world-over, and there are nearly 72 million patients with diabetes in Middle East & North Africa (MENA) region with United Arab Emirates having nearly a million of them.1 The most common type of DM is type 2 DM (nearly 90%) with impaired insulin secretion and usually associated with resistance to insulin actions, while others include gestational diabetes, DM secondary to pancreatic injury, immune mediated type 1 DM and monogenic diabetes. Monogenic diabetes encompasses previously termed maturity onset diabetes of the young as well as neonatal and mitochondrial disease all resulting from single gene defect. The prevalence of Monogenic Diabetes in European and North American population (mainly Caucasians) is 1/10,000 among adults, but for glucokinase (GCK) variant the prevalence can be as high as 1/1000. The prevalence of Monogenic Diabetes / MODY in Middle East population is not known with only two studies of more than 50 patients is Israel and Jordan mainly on GCK subtype. At present over 80% of Monogenic Diabetes patient are misdiagnosed and treated as either Type 1 or Type 2 diabetes mellitus. The commonest forms of treatment-requiring MODY are HNF4-alpha and HNF1-alpha, which do not necessarily require insulin, hence correct diagnosis can be life changing of these patients. There is MODY risk calculator developed by Exeter University that helps predict the presence of Monogenic diabetes but it is validated for Caucasian population only with no data on Emirati population. There are no studies at present on either assessing the presence of MODY in United Arab Emirates population or on identifying MODY patients who are already misdiagnosed with other forms of diabetes.

The aim of this study to assess the presence of common forms of Monogenic diabetes by genetic testing in susceptible adolescents/adults (based on MODY calculator risk factors & antibody testing) who are already diagnosed with Diabetes Mellitus (either type 1 or Type 2)

Objective:

Primary:

To assess the frequency of MODY monogenic diabetes (commonest subtypes) among patients already labelled as Type 1 or Type 2 Diabetes (who have negative autoimmunity, lack of significant ketosis and either family history of diabetes in one parent or BMI<40).

Secondary:

* To assess the validity of MODY risk calculator for prediction of monogenic diabetes in Emirati patients
* To assess the validity of Insulin antibodies in ruling out monogenic diabetes
* To assess the validity of C-peptide activity level in differentiating type 1 diabetes from type 2 diabetes and monogenic diabetes

Data Collection:

The paediatric and adult diabetes clinics in Tawam Hospital Diabetes clinics and clinicians therein will be contacted and any patient meeting the above-mentioned selection criteria will be identified. An informed consent will take from patient and/or parent/guardian explaining the risks and benefits of the study. The patient without insulin antibody testing will undergo testing and only those patients who have negative antibodies will undergo C-peptide activity level (either non-stimulated serum C-peptide or 2-hour post prandial urinary C-peptide creatinine ratio) and only those with absent/reduced C-peptide levels will be excluded. Demographic details and clinical parameters like BMI, duration of diabetes, treatment history and co-morbidities will be obtained. The patient's routine diabetes related blood tests including (HbA1c, liver function tests, albumin, bilirubin, Prothrombin time, albumin, creatinine) done in the last 3months and demographic data (non-identifiable) will be initially gathered on a data collection sheet which will then be transferred to electronic data in Microsoft Excel sheet and stored on a secure server. The MODY risk score will be calculated using the published formula (available at website https://www.diabetesgenes.org/exeter-diabetes-app/ModyCalculator).

The patient will be seen as per routine clinical care and on the next set of blood work additional vials of blood sample will be taken for monogenic testing. No separate venesection or additional visit for the patient will be required. Copy of the monogenic testing will be provided to the clinician in-charge of the patient to help with any clinical decisions.

Confidentiality:

No patient specific identifiable data will be stored in this study. All other data stored will be on United Arab Emirates University secure server. The proposal will be sent to the Research and Ethics committee Tawam for approval as well as to UAEU human ethics committee.

Funding:

There will be funding required for this study for additional testing (including C-peptide activity/antibody testing and genetic testing) as well as for research assistant for 2 years.

Conflict of interest:

None

Financial disclosure:

None

ELIGIBILITY:
Inclusion Criteria:

* Age > 11; both male or female, Emirati patients only
* Diagnosed to have Type 1 or Type 2 Diabetes Mellitus diagnosed before the age of 40 and after the age of 6 months.
* Attended Tawam hospital during the last 1 year.
* All previous antibodies testing being negative.
* Absence of ketoacidosis / significant ketosis in the past medical records

Exclusion Criteria:

* BMI of 40 or above (class 3 / severe obesity)
* History of Secondary diabetes (e.g. Diabetes following pancreatitis)
* Absent/Decreased C-peptide activity suggestive of Type 1 Diabetes

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To see how many patient with diabetes diagnosed at early age with features not suggestive of type 1 or type 2 are found to have MODY monogenic diabetes (commonest subtypes) among young Emirati patients | 24 months
  To assess the frequency of MODY monogenic diabetes (commonest subtypes) among patients already labelled as Type 1 or Type 2 Diabetes (who have negative autoimmunity, lack of significant ketosis and either family history of diabetes in one parent or BMI<40).

SECONDARY OUTCOMES:
To compare the value of MODY risk calculator and genetic testing outcome in Emirati patients | 24 months
  To assess the validity of MODY risk calculator for prediction of monogenic diabetes in Emirati patients
To see if C-peptide activity helps in differentiating monogenic diabetes from type 1 | 24 months
  To assess the validity of C-peptide activity level in differentiating type 1 diabetes from type 2 diabetes and monogenic diabetes
To find out the antibodies present in young patient with diabetes and if they are helpful in ruling out monogenic diabetes | 24 months
  To assess the validity of Insulin antibodies (anti-GAD65, IAA2, Anti-Zn8) in ruling out monogenic diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Agha, Principal Investigator — United Arab Emirates University, College of Medicine & Health Sciences

IPD SHARING:
Plan to Share IPD: No
At the end of the study datasheet with clinical and biochemical parameters including antibody, MODY risk calculation, C-peptide activity and genetic testing results (with no personal identifiable information) could be shared.

REFERENCES:
- [Background] Taneera J, Mussa B, Saber-Ayad M, Dhaiban S, Aljaibeji H, Sulaiman N. Maturity-Onset Diabetes of the Young: An Overview with Focus on the Middle East. Curr Mol Med. 2017;17(8):549-562. doi: 10.2174/1566524018666180222121158. PMID 29473506
- [Background] Shields BM, McDonald TJ, Ellard S, Campbell MJ, Hyde C, Hattersley AT. The development and validation of a clinical prediction model to determine the probability of MODY in patients with young-onset diabetes. Diabetologia. 2012 May;55(5):1265-72. doi: 10.1007/s00125-011-2418-8. Epub 2012 Jan 5. PMID 22218698
- [Background] Hattersley AT, Patel KA. Precision diabetes: learning from monogenic diabetes. Diabetologia. 2017 May;60(5):769-777. doi: 10.1007/s00125-017-4226-2. Epub 2017 Mar 17. PMID 28314945